CLINICAL TRIAL: NCT03152032
Title: Employment Outcomes After In-House Vocational Training Programs for Individuals With Chronic Psychiatric Disorders
Brief Title: Employment Outcomes After Vocational Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TsaoTun Psychiatric Center, Department of Health, Taiwan (Other)
Responsible Party: Principal Investigator, Eric J. Hwang, Clinical research mentor, TsaoTun Psychiatric Center, Department of Health, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EH32469
Record Dates: First submitted 2017-05-08; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Schizophrenia and Related Disorders; Bipolar and Related Disorders
Keywords: employment service; vocational counseling; employment outcome; schizophrenia; bipolar; occupational therapy in mental health
MeSH Terms: conditions — Schizophrenia; Bipolar and Related Disorders

STUDY DESIGN:
Intervention Model Description: All study participants attended the vocational training program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In-House Vocational Training Programs (Experimental): The In-House Vocational Training Programs were government-funded services offered to newly discharged inpatients or current outpatients with chronic psychiatric disorders in four regional psychiatric hospitals of Taiwan. The programs emphasized the utilization of the hospitals' existing spaces, facilities and manpower alongside the community sources to train participants in various job options including bakery training, culinary skill, barista training, computer data processing, auto wash and detailing, janitorial training, and wash and fold laundry service. Each program was staffed with occupational therapists and paid or volunteer job coaches, along with cross-disciplinary support from psychiatrists, psychologists, social workers, nurses, vocational specialists or others.
  Interventions: Behavioral: In-House Vocational Training Programs

INTERVENTIONS:
Behavioral: In-House Vocational Training Programs — At the beginning of the IHVT programs, the job placement for each participant was determined jointly by the participant's interest, the demands of local job markets and the team evaluation. The programs covered 6 to 10 months in length, 5 days a week and 4 to 6 hours a day. The programs contained three sessions: (a) the work-related behavior training session, such as proper appearance, communication and self assertion, and workplace social skills, (b) the on-the-job skill training session where participants gained job-specific training and interventions from job coaches and occupational therapists, and (c) the life balance counseling session including individual and group counseling that aimed to enhance the participants' ability to tackle potential hardships and barriers to work.
  Other Names: IHVT Programs

SUMMARY:
This multicenter retrospective cohort study examined the employment outcomes of the innovative in-house vocational training (IHVT) programs for individuals with chronic psychiatric disorders (CPD) and explored the program parameters significantly predictive of the outcomes. The IHVT programs were government-funded services offered to newly discharged inpatients or current outpatients with chronic psychiatric disorders (CPD) in four regional psychiatric hospitals of Taiwan. Each program was staffed with occupational therapists and paid or volunteer job coaches, along with cross-disciplinary support from psychiatrists, psychologists, social workers, nurses, vocational specialists or others. Data were retrieved from 323 participants with CPD who completed the IHVT and the 1st-, 3rd-, and 6th-month follow-up interviews. The employment outcomes examined were the participants' employment rates at the 1st-, 3rd-, and 6th-month post-training as well as their sustainability of employment during the 6 months post-training.

DETAILED DESCRIPTION:
The Purpose of the Study

This study aimed to explore the employment outcomes of the In-House Vocational Training ( IHVT) programs by examining participants' employment rates at the 1st-, 3rd-, and 6th-month follow-ups as well as their overall sustainability of employment during the first 6 months post-training. In addition, we attempted to determine the program parameters (e.g., pre-training screening and evaluation, therapist training and experience, cross-disciplinary initiative, and counseling service) that had a significantly positive effect on the employment outcomes.

Research Design

This was a multicenter retrospective cohort study utilizing data retrieved from the files of the IHVT participants in four regional psychiatric hospitals of Taiwan.

Recruitment of Participants

The retrospective cohort study utilized data of 323 participants from four regional psychiatric hospitals in Taiwan who met the following criteria: (a) being 18 year-old or older, (b) having a diagnosis of DSM-V psychiatric disorder for a minimum of 12 months, (c) being a newly discharged inpatient (< 3 months) or current outpatient of one of the aforementioned psychiatric hospitals in Taiwan, (d) having completed the entire IHVT program described below as well as the 1st, 3rd-, and 6th-month follow-up interviews, and (d) having signed participant informed consent. The Institution Review Board and Research Ethics Committee of the project sponsor (Tsaotun Psychiatric Center, Ministry of Health and Welfare, Nantou County, Taiwan) approved the project proposal and oversaw the procedures of participant recruitment, intervention (training) programs, and data collection and analyses.

Intervention: In-House Vocational Training Programs (IHVT)

The IHVT programs were government-funded services offered to newly discharged inpatients or current outpatients with chronic psychiatric disorders (CPD) in four regional psychiatric hospitals of Taiwan. Each program was staffed with occupational therapists (including the program direct, case managers and on-site therapists) and paid or volunteer job coaches, along with cross-disciplinary support from psychiatrists, psychologists, social workers, nurses, vocational specialists or others. The programs emphasized the utilization of the hospitals' existing spaces, facilities and manpower alongside the community sources and networks to train their participants in a range of job options including bakery training, culinary skill, barista training, computer data processing, auto wash and detailing, janitorial training, and wash and fold laundry service. The job placement for each participant was determined jointly by the participant's interest, the demands of local job markets and the results of evaluation by the case manager or a cross-disciplinary team. The IHVT programs generally covered 6 to 10 months in length (varying with the job options), 5 days a week and 4 to 6 hours a day.

The IHVT programs contained three sessions throughout the entire course of training: (a) the work-related behavior training session, (b) the on-the-job skill training session, and (c) the life balance counseling session. The work-related behavior training session included a rich array of lectures and discussion, group activities and presentations, and take-home assignments. The topics may include, but are not limited to, proper appearance and attire; punctuality, attendance and responsibility; communication and self assertion; engagement, concentration, and work completion; workplace social skills and etiquette; problem solving and conflict resolution; and job searching and interview skills. The on-the-job skill training session took place in the hospitals' facilities or affiliations, such as the hospitals' bakeries, coffee shops, restaurants, cafeterias, offices, janitorial departments, laundry facilities and car wash/detailing workshops. These facilities were all housed in the hospitals or their vicinity and many were open to the public (e.g., bakeries, coffee shops, restaurants, and car wash/detailing workshops). It was a half- or full-day unpaid internship where the participants gained job-specific training and hands-on experience from the job coaches and, at the same time, received necessary supervision, guidance and interventions from the on-site occupational therapists. Moreover, the life balance counseling session consisted of individual and group counseling that aimed to enhance the participants' ability to tackle potential hardships and barriers to work. Stress management and relaxation techniques, coping strategies, work and leisure, time management, medication issues, self-advocacy, and community outreach and resources were the common areas for counseling offered by occupational therapists (case managers) or cross-disciplinary initiatives (e.g., psychiatrists, psychologists, social workers, nurses or other). Finally, post-training vocational counseling services provided by the IHVT case manager or other vocational specialists in community settings were also available to the participants so as to continuously promote their employment capacity. Of note, while incorporating all the essential sessions and components of the IHVP, the four participating hospitals demonstrated variations in some program parameters (e.g., length, staffing, job training options, post-training counseling services) due to their inherent differences in infrastructure, manpower and resources.

Research Variables

Outcome/dependent variables: The outcome variables of this study were employment rates and employment sustainability. Employment rates were the percentages of participants who were employed at the 1st-, 3rd-, and 6th-month follow-up interviews, respectively. For the purpose of this study, participants were deemed "employed" if they had a full-time paid job (a workload of 30 hours or more per week) in any of the following work placements: sheltered, supported, or competitive employment. In turn, the employment sustainability during the first 6 months post-training was graded into five levels: (a) high sustainability (5 points), (b) medium sustainability (4 points), (c) medium low sustainability (3 points), (d) low sustainability (2 points), and (e) very low sustainability (1 point). The detailed definitions of the employment sustainability levels will be described in Results.

Independent variables: Independent variables were the related program parameters that might significantly correlate with participants' employment outcomes. A total of 8 program parameters were identified: (a) participant's pre-training screening/evaluation, (b) therapist's obtaining a specific job certification/licensure, (c) case manager's length of time in practice, (d) case manager's experience in community settings, (e) cross-disciplinary support for life balance counseling, (f) the amount of life balance counseling (hours per week), (g) type of professionals available for post-training vocational counseling, and (h) time parameters post-training (1st, 3rd or 6th month). The detailed definitions of these program parameters will be described in Results.

Control variables. In order to determine which of the aforementioned program parameters (independent variables) could significantly support participants' employment outcomes, we treated "client factors" as control variables to offset their potential confounding effects on the outcomes. These client factors included participants' demographics (i.e., gender, educational attainment, marital status, and age), diagnostic characteristics (i.e., major diagnosis, age of onset, and length of time since onset) and functional levels (i.e., hand function, attention span, and activities of daily living [ADL] skill). The instruments used to measure participants' functional levels are described below.

Instrumentation

Data regarding participants' functional levels were collected through Chu's Occupational Assessment Inventory that consists of Hand Dexterity Test, Attention Test, and Activities of Daily Living (ADL) Test - 2nd ed. These tests were purposefully developed and validated for use with individuals diagnosed with psychiatric disorders. The administration of Chu's Occupational Assessment Inventory has been a routine, standard evaluation procedure in many psychiatric occupational therapy settings in Taiwan. Norms for the three tests were established through the national samples of Taiwan. Functional levels assessed through each of the three tests were calibrated into: 5 - Good, 4 - Fair, 3 - Mild Impairment, 2 - Moderate Impairment, 1 - Severe Impairment, and 0 - Very Severe Impairment. Reliability and validity of the three tests have been well supported in previous studies.

Data Analysis

Data were analyzed using IBM SPSS Statistics 22. Descriptive statistics and frequency analysis were first conducted to summarize the data sets. Univariate analyses for the categorical independent variable (employed or unemployed) including Chi-square test and simple logistic regression, and univariate analyses for the continuous dependent variable (employment sustainability) including one-way analysis of variance (ANOVA) and correlation (Pearson's r) were used to preselect independent variables (program parameters) and control variables (client factors) that could have an effect on participants' employment outcomes. Subsequently, we performed the generalized estimating equation (GEE) to analyze our 1st-, 3rd- and 6th-month longitudinal employment data with the preselected independent variables offset by the control variables to conclude the program parameters significantly predictive of participants' employment rates and employment sustainability, respectively.

Research Questions

1. What were the participants' employment rates at the 1st-, 3rd-, and 6th-month follow-ups post training, respectively?
2. What was the participants' overall sustainability of employment during the first 6 months post-training?
3. What were the program parameters (e.g., pre-training screening and evaluation, therapist training and experience, cross-disciplinary initiative, and counseling service) that had a significantly positive effect on the employment rates and the sustainability of employment?

ELIGIBILITY:
Inclusion Criteria:

* 18 year-old or older
* a diagnosis of DSM-V psychiatric disorder for a minimum of 12 months
* a newly discharged inpatient (< 3 months) or current outpatient of one of the four participating psychiatric hospitals in Taiwan
* completed the entire IHVT program
* completed the 1st, 3rd-, and 6th-month follow-up employment interviews
* signed participant informed consent

Exclusion Criteria:

* Participants who did not fully complete the IHVT program
* Participants who missed any of the 1st, 3rd-, and 6th-month follow-up employment interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
The employment rate at the 1st-month post-training interview | 1st-month post-training
  The employment rate was the percentages of participants who were employed at the 1st-month post-training follow-up interview. In this study, participants were deemed "employed" if they had a full-time paid job (a workload of 30 hours or more per week) in any of the following work placements: sheltered, supported, or competitive employment.
The employment rate at the 3rd-month post-training interview | 3rd-month post-training
  The employment rate was the percentages of participants who were employed at the 3rd-month post-training follow-up interview. In this study, participants were deemed "employed" if they had a full-time paid job (a workload of 30 hours or more per week) in any of the following work placements: sheltered, supported, or competitive employment.
The employment rate at the 6th-month post-training interview | 6th-month post-training
  The employment rate was the percentages of participants who were employed at the 6th-month post-training follow-up interview. In this study, participants were deemed "employed" if they had a full-time paid job (a workload of 30 hours or more per week) in any of the following work placements: sheltered, supported, or competitive employment.

SECONDARY OUTCOMES:
Employment sustainability during the first 6 months post-training | the first 6 months post-training
  Employment sustainability during the first 6 months post-training was graded into five levels: (a) high sustainability (employed throughout the 1st, 3rd, and 6th months post-training.), (b) medium sustainability (employed during 1st and 3rd months or 3rd and 6th months), (c) medium low sustainability (employed in 1st and 6th months), (d) low sustainability (employed only in 1st, 3rd, or 6th month), and (e) very low sustainability (not employed throughout the 1st, 3rd, and 6th months post-training).

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ling Lee, MS, Principal Investigator — Tsaotun Psychiatric Center, Nantou County, Taiwan

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan.

REFERENCES:
- [Background] Arbesman M, Logsdon DW. Occupational therapy interventions for employment and education for adults with serious mental illness: a systematic review. Am J Occup Ther. 2011 May-Jun;65(3):238-46. doi: 10.5014/ajot.2011.001289. PMID 21675329
- [Background] Bond GR, Drake RE, Becker DR. An update on randomized controlled trials of evidence-based supported employment. Psychiatr Rehabil J. 2008 Spring;31(4):280-90. doi: 10.2975/31.4.2008.280.290. PMID 18407876
- [Background] Chuang WF, Hwang E, Lee HL, Wu SL. An in-house prevocational training program for newly discharged psychiatric inpatients: exploring its employment outcomes and the predictive factors. Occup Ther Int. 2015 Jun;22(2):94-103. doi: 10.1002/oti.1388. Epub 2015 Mar 16. PMID 25783143
- [Background] Jang Y, Wang YT, Lin MH. Factors affecting employment outcomes for people with disabilities who received Disability Employment Services in Taiwan. J Occup Rehabil. 2014 Mar;24(1):11-21. doi: 10.1007/s10926-013-9433-1. PMID 23512347
- [Background] Waghorn G, Dias S, Gladman B, Harris M, Saha S. A multi-site randomised controlled trial of evidence-based supported employment for adults with severe and persistent mental illness. Aust Occup Ther J. 2014 Dec;61(6):424-36. doi: 10.1111/1440-1630.12148. Epub 2014 Oct 4. PMID 25284162
- [Derived] Lee HL, Hwang EJ, Wu SL, Tu WM, Wang MH, Chan F. Employment Outcomes After Vocational Training for People With Chronic Psychiatric Disorders: A Multicenter Study. Am J Occup Ther. 2018 Sep/Oct;72(5):7205195010p1-7205195010p9. doi: 10.5014/ajot.2018.028621. PMID 30157009